CLINICAL TRIAL: NCT05299385
Title: Multicenter, Prospective, Comparative, Randomized, Single Blind, Superior, Pivotal Study to Evaluate the Clinical Effectiveness and Safety of Respiratory Rehabilitation Software 'Redpill Breath' Compared to the Manual Rehabilitation Management(COPD, Asthma, Lung Cancer, Etc.)
Brief Title: The Study for Evaluating the Clinical Effectiveness and Safety of Respiratory Rehabilitation Software 'Redpill Breath'(COPD, Asthma, Lung Cancer, Etc.)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lifesemantics Corp. (Industry)
Collaborators: Asan Medical Center (Other); KangWon National University Hospital (Other); SMG-SNU Boramae Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LFSPMR-01
Record Dates: First submitted 2022-01-11; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Respiratory System Disease; Chronic Obstructive Pulmonary Disease; Asthma Copd; Lung Cancer; Lung Diseases; Pulmonary Rehabilitation; Respiratory Rehabilitation; Home Based Rehabilitation; Mobile Application; Rehabilitation
Keywords: DTx; Digital therapeutics; PR; COPD
MeSH Terms: conditions — Respiratory Tract Diseases; Pulmonary Disease, Chronic Obstructive; Lung Neoplasms; Lung Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Comparator (Active Comparator): The investigator provide conventional-treatment to subjects when distributing respiratory rehabilitation education leaflets, Investigators explain the leaflets and self-practice until the subjects fully understand them. Compactor conducts respiratory rehabilitation treatment for 12 weeks according to the following procedures at home
  ☞ The investigator shall contact the subject every two weeks during the respiratory rehabilitation period and encourage them to perform respiratory rehabilitation treatment according to the assigned group. Subjects perform respiratory rehabilitation exercises at home.
  They have to visit hospital at 8 weeks (visit 3) and 12 weeks (visit 4) and then examine the factor of the outcome measure following the clinical protocol
  Interventions: Behavioral: Conventional rehabilition treatment(e.g leaflet) educated by hospital
- Experimental treatment (Experimental): Subjects install software as a medical device for clinical trials on smart-phones, so that the subject can perform respiratory rehabilitation treatment at home.
  Respiratory rehabilitation treatment for 12 weeks
  ☞ Respiratory rehabilitation treatment using a mobile-based software, consists of aerobic exercise and anaerobic exercise, and the subject performs themselves
  They have to visit hospital at 8 weeks (visit 3) and 12 weeks (visit 4) and then examine the factor of the outcome measure following the clinical protocol
  Interventions: Device: Digital treatment based on Respiratory Rehabilitation Software

INTERVENTIONS:
Behavioral: Conventional rehabilition treatment(e.g leaflet) educated by hospital — Active Comparator: subjects who are trained in accordance with the conventional manual treatment of Respiratory rehabilitation in the clinical institution and taking care home-based management.
  The manual contents
  * method of the conventional rehabilitation treatment
  * intensity for aerobic exercise and anaerobic exercise
  Other Names: the conventional rehabilitation treatment
  Arms: Comparator
Device: Digital treatment based on Respiratory Rehabilitation Software — Experimental: subjects who use the software as a home-based Digital Respiratory Rehabilitation software
  It is intended for subjects who are prescribed a respiratory rehabilitation exercise to improve their physical condition. The software also helps them to do self-rehabilitation exercise.
  Other Names: Respiratory Rehabilitation Software
  Arms: Experimental treatment

SUMMARY:
The purpose of the study is to prove the clinical superiority of respiratory rehabilitation software "Redpill Breath" and evaluate the clinical improvement effect by 6-minute walk test of the software, compared to the manual rehabilitation management for those who need respiratory rehabilitation(COPD, Asthma, Lung Cancer, etc.)

ELIGIBILITY:
Inclusion Criteria:

1. 19 to 80 years-old
2. Subject who has difficulty in respiratory symptoms and routine with the criteria as below 1) mMRC(modified Medical Research Council Dyspnea Scale) 1 point at least 2) In accordance with Pulmonary function test(PFT/LET/EEG) examined, if there is in one of the following cases as below [a lung cancer patient] (FVC or FEV1 < 80%), [No lung cancer patient] (Post-bronchodilator FEV1/FVC < 0.7) and (Post-bronchodilator FEV1 < 80%)
3. Subject with an Android smartphone (OS 8.0 or higher, internal memory (HDD) of 32GB or higher) or iPhone (iOS 13.0 or higher, internal memory (HDD of 32GB or higher)
4. Subject who can use effectively smartphone and mobile software
5. Subject who brings their smartphone for a walking test during 12 weeks of the clinical trial.
6. Subject who makes the decision voluntarily for participating in the clinical trial and to write their signature to the consent of subject's explanation.
7. Subject who complies with the clinical protocol

Exclusion Criteria:

1. Subject who has respiratory distress syndrome, caused by a kind of Neuromuscular disease, Spinal cord injury, Thoracic deformation, etc.
2. Subject who participate in respiratory rehabilitation treatment within 6 months of the screening date
3. Subject who undergoes respiratory-related symptoms deteriorate within 2 weeks of the screening date to the point where they need additional antibiotics or steroids
4. Subject who has an unstable cardiovascular disease (unstable angina pectoris, Acute myocardial infarction, severe coarctation of aorta, etc.)
5. a pulmonary arterial hypertension subject
6. Subject prescribed physical(e.g. lower-leg joint surgery, neurological limitation) or cognitive factors(e.g. psychical disorder)
7. Pregnant or lactating women
8. Subject who is unable to read text and tough to communicate
9. Subject who has participated in other clinical trials within 90 days of the screening date or participating in other clinical trials.
10. Subject who is determined to inappropriate to perform this study according to clinical research associate's opinion(e.g if someone has a bearing on the result of the clinical trial ethically or clinically)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2022-03-28 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
The 6-minute walking distance (6 minute walking distance, 6MWD) change amount(in meters) at 12 weeks after respiratory rehabilitation compared to the baseline. | 12 weeks
  the primary efficacy variable is the change of respiratory function parameters as a 6-minute walking distance(6MWT) in meters(m) at V4 compared with the baseline(V2). The value of 6MWD at V2 adjust as the value of covariate for statistical significance between the groups.

SECONDARY OUTCOMES:
The 6-minute walking distance (6 minute walking distance, 6MWD) change amount(in meters) at 8 weeks after respiratory rehabilitation compared to the baseline. | 8 weeks
  the efficacy variable is the change of respiratory function parameters (6MWT) at V3 compared with the baseline(V2). Statistical significance is tested through the Independent two-sample-test or the Wilcoxon rank sum test. it will be evaluated separately from the primary outcome(6MWD at 12 weeks)
The amount of change in the modified medical ressearch council Dyspnea scale (mMRC) scores at 8 and 12 weeks after respiratory rehabilitation compared to the baseline. | 8 and 12 weeks
  the efficacy variable is the change of respiratory function parameter by modified medical research council Dyspnea scale(mMRC) scores at V3 and V4 compared with the baseline(V2). the total score ranges from 0 to 4, The higher score means more severe symptoms. Statistical significance of changes within each group is tested by the Paired -test or Wilcoxon signed rank test.
The amount of change in the Structures Respiratory Questionnaire (SGRQ) score at 8 and 12 weeks after respiratory rehabilitation compared to the baseline. | 8 and 12 weeks
  the efficacy variable is the change of respiratory function scores(Structures Respiratory Questionnaire, SGRQ) at V3 and V4 compared with the baseline(V2). Scores range from 0 to 100, with higher scores indicating more limitations. Statistical significance of changes within each group is tested by the Paired -test or Wilcoxon signed rank test.
The amount of change in the Hospital Anxiety and Depression Scale (HADS) at 8 and 12 weeks after respiratory rehabilitation compared to the baseline. | 8 and 12 weeks
  the efficacy variable is the change of respiratory function scores(Hospital Anxiety and Depression Scale, HADS) at V3 and V4 compared with the baseline(V2). Scores range from 0 to 21, with the higher score indicating the more depressed and anxious. Statistical significance of changes within each group is tested by the Paired -test or Wilcoxon signed rank test.
The amount of change in the average number of daily steps per week during the respiratory rehabilitation management period (number of times) | per week for 12weeks
  the efficacy variable is the daily step count detection using medical device for 12 weeks. Statistical significance of changes within each group is tested by the Paired -test or Wilcoxon signed rank test.
The number of times in the use of medical support (days of hospitalization) | 12 weeks
  the efficacy variable is number of days of hospitalization for 12 weeks compared with the baseline(V2). Statistical significance of changes within each group is tested by the Paired -test or Wilcoxon signed rank test.
The number of times in the use of medical support (days of emergency room visits) | 12 weeks
  the efficacy variable is number of days of hospitalization, number of days of emergency room visits for 12 weeks compared with the baseline(V2). Statistical significance of changes within each group is tested by the Paired -test or Wilcoxon signed rank test.
Abnormal case (safety evaluation variable) | 8 and 12 weeks
  The analysis of abnormal case analyzes all abnormal cases(TEAE) that occurre after the application of medical devices for clinical trials.
  Descriptive statistics(the number of subjects, incidence, and occurrence of coded adverse events) are presented by group. Treatment Emergency Adverse Event (TEAE), Adverse Device Effect (ADE), and Serious Adverse Event (SAE), and the difference in ratio between groups analyzes through Chi-square test or Fisher's exact test. The factors are coded according to SOC and PT using MedDRA. In addition, a detailed list is presented for individual subjects who have experienced significant abnormalities.
Patient Global Assessment (PGA) evaluation for 12 weeks after respiratory rehabilitation management | 12 weeks
  the scores of experimental group's Patient Global Assessment (PGA) evaluation using medical device for 12 weeks. PGA is assessed by a single question ranged from 0 to 10. the higher score means the greater patient's satisfaction.
Evaluation of the number of treatments during the respiratory rehabilitation management period (number of times) | 12 weeks
  the experimental group's the number of treatments, using medical device for 12 weeks represents descriptive statistics (number of subjects, average, standard deviation, median, minimum, and maximum value)

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Kangwon National University Hospital, Chuncheon
  - Asan Medical Center, Seoul
  - Kangwon National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No